CLINICAL TRIAL: NCT04132349
Title: The Effectiveness and Safety of Ulipristal Acetate in Women With Symptomatic Uterine Fibroid
Brief Title: Ulipristal Acetate in Symptomatic Uterine Fibroid
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Ulipristal Acetate was recalled
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS/BVMD/19/12
Record Dates: First submitted 2019-10-15; First posted 2019-10-18 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Uterine Fibroid; Heavy Menstrual Bleeding
Keywords: Ulipristal Acetate
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — ulipristal acetate

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ullipristal Acetate (Experimental): Women with symptomatic uterine fibroids will be treated with 5 mg UPA / day in 3 months
  Interventions: Drug: Ulipristal Acetate 5 mg

INTERVENTIONS:
Drug: Ulipristal Acetate 5 mg — Ulipristal acetate (from Cenexi manufacturer, France) at daily dose of 5mg in 3 consecutive months course
  Other Names: Esmya

SUMMARY:
This study evaluates the effectiveness and safety of ulipristal acetae (UPA) in women with symptomatic uterine fibroids. Those who fulfilled inclusion/exclusion criteria will be treated UPA at daily dose of 5mg.

DETAILED DESCRIPTION:
There is increasing evidence approving role of medical therapy in treatment of symptomatic uterine fibroid, in the context of women's desire to preserve fertility or not to undergo operation.

Among these hormonal therapies, ulipristal acetate (UPA) is an orally administered selective progesterone receptor modulator commonly prescribed for treatment of uterine fibroid. This agent acts on causing apoptosis of the muscle cells inside the tumor and reducing the tumor matrix in case of uterine fibroid.

UPA at daily dose of 5 mg has been shown to decrease menstrual blood loss and reduce tumor size after 13 consecutive weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-48
* Regular cycle of 22-35 days interval and FSH <=20 mUI/mL.
* >=1 uterine fibroid of 3<= d < 10cm (regardless of location), diagnosed by transvaginal ultrasound.
* Heavy menstrual bleeding (blood loss >80ml/cycle).
* Uterine size < 16 weeks of GA on clinical examination.
* Agree to participate in the study.

Exclusion Criteria:

* Previous or current treatment of uterus, cervix, ovarian or breast cancer.
* Previous endometrial ablation or uterine artery embolization.
* Abnormal PAP's smear result within 12 months prior to recruitment.
* Endometrial hyperplasia within 6 months prior to recruitment.
* Uterine polyp >2cm.
* Ovarian cysts 4cm diagnosed by transvaginal ultrasound.
* Severe anemia (Hb 6 g/dl) or indication for blood transfusion.
* Coagulation disorder indicated for treatment.
* Increased liver enzyme level of twofold or more than normal upper limit.
* Previous use of SPRM.
* Treatment of systemic progestin or intrauterine device or hormonal contraception within 2 months, or use of GnRH analogue within 5 months prior to recruitment.
* Current use of acetylsalicylic acid, mefenamic acid, anticoagulation agents, antifibrinolysis agents, or systemic corticoid

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Amenorrhea | from first dose to the end of 3 consecutive months of treatment course
  Percentage of subjects achieve amenorrhea at the end of treatment. Amenorrhea is defined of 35 consecutive non-bleeding days, in which spotting is accepted.

SECONDARY OUTCOMES:
time from treatment to amenorrhea | from first dose to the end of 3 consecutive months of treatment course
  the number of days from treatment initiation to the date that the subject has achieved amenorrhea.
uterine fibroid size change | from first dose to the end of 3 consecutive months of treatment course
  the total volume of the 3 largest uterine fibroids will be measured. Uterine fibroid size change will be calculated by percentage of the figure at the end of treatment in comparison to at baseline.
pelvic pain control | from first dose to the end of 3 consecutive months of treatment course
  Pelvic pain assessed by visual analogue score (VAS). The minimum score is 0, which means no pain at all. The maximum score is 10, which means unbearable pain. Higher scores mean worse outcome.
adverse events | from first dose to the end of 3 consecutive months of treatment course, and the end of 3 months follow-up without treatment
  Percentage of participants have adverse events. Adverse events are defined as any undesirable experience occurring to a subject during a clinical trial, whether or not considered related to the intervention
Uterine fibroid symptom and health - related quality of life score change | from first dose to the end of 3 consecutive months of treatment course
  Uterine Fibroid symptom and health - related quality of life questionnaire (UFS-QOL) consists of 37 questions to assess symptoms of uterine fibroid and their impacts on women's quality of life. Each answer is scored from 1 to 5, in which 1 equals not at all and 5 equals all of the time. The minimum score is 0 and the maximum score is 185. Higher scores mean worse outcome.
Abnormal endometrial features and thickness | from first dose to the end of 3 consecutive months of treatment course
  Endometrial thickness is assessed via transvaginal ultrasound every month after initiation of treatment. Endometrial biopsy is performed at baseline and at the end of treatment.
abnormal liver function test findings | from first dose to the end of 3 consecutive months of treatment course
  Liver enzym (AST, ALT) is assessed every month after initiation of treatment. A two-fold or more increase in level of liver enzym is abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Dang Q Vinh, MD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- My Duc Hospital, Ho Chi Minh City, Vietnam